CLINICAL TRIAL: NCT03370627
Title: Effect of Monoclonal Anti-cd303 on the Inhibition of Type I Interferon Secretion in the Peripheral Blood of Patients With Autoimmune Diseases
Brief Title: Effect of Anti-CD303 Antibodies in Autoimmune Diseases
Acronym: ANTI-CD303
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017_23; 2017_A02244-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Immune Disease
Keywords: Autoimmune Diseases; Plasmacytoid Dendritic Cells; Type I Interferons; Antibodies; Anti-CD303
MeSH Terms: conditions — Immune System Diseases; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient (Experimental)
  Interventions: Biological: Monoclonal anti-cd303 antibody

INTERVENTIONS:
Biological: Monoclonal anti-cd303 antibody — Addition of monoclonal anti CD303 antibodies or not (control) on 2 blood samples of the same patient, to which 10 μl of CpG (20 μg / ml) are added in order to activate plasmacytoid Dendritic Cells and to induce the secretion of Type I interferons.

SUMMARY:
The pathogenic role of type I interferons (IFNs) in the development of different autoimmune diseases has been extensively described in the literature. Since plasmacytoid dendritic cells (pDCs) are the main source of type I IFNs, there is evidence of the involvement of pDCs in autoimmune diseases. The CD303 surface protein (also called BDCA-2) is specifically expressed by the pDCs.

The hypothesis leading to the realization of this study is to observe, in vitro, an inhibition of the secretion of the type I IFNs by pDCs in the peripheral blood in patients with autoimmune disease, thanks to the action of the anti-CD303 antibody Developed by the LFB Group, which could reduce the inflammatory response and improve patients with autoimmune disease

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand the requirements of the study, provide written informed consent, and comply with the study data collection procedures
* Patient followed in the department of internal medicine of CHU Lille
* Patient with one of the following autoimmune disease, defined according to international criteria: systemic lupus erythematosus, systemic sclerosis, Gougerot-Sjögren syndrome and idiopathic thrombocytopenic purpura
* Being socially insured

Exclusion Criteria:

* Overlapping syndrome with another autoimmune disease
* Age ≤18 years
* Pregnant or nursing women
* People in emergencies
* Person incapable of consent
* Persons deprived of liberty
* Persons without social security cover

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
in vitro determination of the level of type I interferons by immunoenzymatic ELISA method. | Baseline

SECONDARY OUTCOMES:
in vitro determination of the level of type I interferons by immunoassay ELISA (by type of MIA) | Baseline
in vitro determination of the level of type I interferons by ELISA immunoassay method in patients treated or not with immunosuppressive or immunomodulatory treatment. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: David Launay, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France